CLINICAL TRIAL: NCT04383015
Title: Carbohydrate Requirements for Prolonged, Fasted Exercise With and Without Basal Rate Reductions in Individuals With Type 1 Diabetes on Continuous Subcutaneous Insulin Infusion
Brief Title: Carbohydrate and Insulin Requirements During Prolonged Fasted Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Insulet Corporation (Industry)
Responsible Party: Principal Investigator, Michael Riddell, Principal Investigator, York University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: e2018-306
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Type 1 Diabetes
Keywords: Physical Activity; Exercise; Carbohydrates; Hypoglycemia; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Patients with type 1 diabetes on insulin pump therapy will remain on their usual insulin regimen. However, we are testing percent basal rate reductions during exercise (50 percent reduction) with or without carbohydrate feeding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate (CHO)-only (Other): Carbohydrate dose of 0.3g/kg/hr given every 30 minutes of exercise if blood glucose is in range with usual basal insulin infusion
  Interventions: Other: Exercise strategies
- 50 Percent Basal Rate Reduction (BRR) (Other): A 50 percent basal rate reduction set 90-minutes pre-exercise and throughout exercise
  Interventions: Other: Exercise strategies
- Combo (Other): The combination of a 50 percent basal rate reduction and carbohydrate dose of 0.3g/kg/hr (given every 30 minutes) both at exercise onset
  Interventions: Other: Exercise strategies

INTERVENTIONS:
Other: Exercise strategies — Strategies for exercise in type 1 diabetes to maintain glucose control

SUMMARY:
The purpose of this study is to compare the time spent in glucose target range (4.0-10.0 mmol/L) during exercise and in recovery using three different management strategies for prolonged aerobic exercise: A) carbohydrate dose of 0.3g/kg/hr; B) A 50 percent basal rate reduction, performed 90-minutes in advance of exercise for the duration of the activity; and C) A 50 percent basal rate reduction, performed at exercise onset, with carbohydrate dose of 0.3g/kg/hr

DETAILED DESCRIPTION:
This project focuses on the effectiveness of various exercise strategies on the time spent in target range during and after aerobic exercise in adults with type 1 diabetes (T1D) on continuous subcutaneous insulin infusion (CSII).

The primary objective of the protocol is to determine if a moderate basal insulin reduction (-50 percent of basal), performed 90-minutes before a 120-minute aerobic exercise session (with 5-minute breaks every 30 minutes of exercise, and a ten minute break mid-exercise), improves the time in target range compared to either a carbohydrate consumption only strategy or insulin reduction (-50 percent) and carbohydrate consumption strategy both performed at the onset of exercise in patients with T1D on CSII therapy. The time in target will be determined for both the exercise period and during a 24-hour window after the end of exercise.

In all three sessions, aerobic exercise (brisk walking) will be performed in the fasted state (minimum 8 hours after the last meal) in the early-morning. The exercise will consist of four 30-minute bouts of walking at 40-50 percent of the participant's pre-determined aerobic capacity, separated by 5-10 minute breaks. The participants exercise intensity will be monitored continuously using heart rate and activity monitors. Blood glucose and blood ketone levels will be monitored throughout exercise.

Each participant will be assigned to a sequence of the three experimental visits through a randomization process. Each exercise session will be separated by at least two days and participants will be expected to complete all sessions within ~ 12 weeks from the time of the baseline/screening visit. Participants will be instructed to apply a new continuous glucose monitor (CGM) sensor between 1-5 days prior, not to perform moderate-to-vigorous exercise 24 hours prior and refrain from caffeine and alcohol 12 hours prior to each study visit. Participants are also instructed not to eat after 2330h the night before arriving to the laboratory and not to give bolus insulin or perform temporary basal rate changes after 0200h on the morning of the exercise visit. Participants are instructed to try to arrive at the laboratory with their blood glucose between 72-270 mg/dL, with no active bolus insulin according to personal CSII device, in the fasted state. If a bolus of insulin was given prior to the exercise session, the session was rescheduled. Females of reproductive capacity performed all three visits in the early follicular phase (days 1-6 of cycle). Participants arrived at the laboratory between 0600h and 1000h. Exercise start time was between 0700h and 1045h, based on participants' choice, and the timing of exercise was kept consistent within participants.

Following each exercise session, the participant will rest for 20-minutes and then leave the laboratory. The participants glucose will be monitored for 24-hours after the standardized exercise. They will also be instructed to perform a standardized basal insulin reduction overnight to help reduce the risk of post-exercise nocturnal hypoglycemia (-20 percent from bedtime for 6 hours).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of presumed autoimmune type 1 diabetes
* Last HbA1c ≤ 9.9 percent
* Age: 17+ years
* Duration of T1D: ≥ 1.5 years
* Using insulin pump therapy: ≥3 months (at least 0.25 units of insulin per kilogram of body mass)
* In good general health with no conditions that could impact the outcome of the trial
* Willing to adhere to the protocol requirements for the duration of the study

Exclusion Criteria:

* Physician diagnosis of active diabetic retinopathy that could be worsened by exercise
* Physician diagnosis of peripheral neuropathy or autonomic neuropathy
* Medications:

  1. Beta-blockers
  2. Agents that affect hepatic glucose production (xanthine derivatives)
  3. Pramlintide
  4. Any other hypoglycemic agent
* Participation in other studies involving the administration of an investigational drug or device during the duration of the current study
* Severe hypoglycemia in the last 3 months, defined as the individual requiring third party assistance or hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Time in glucose target range during exercise intervention | 140 minutes
  The primary outcome measurement is to determine which strategy had the best time in blood glucose target range (4.0-10.0 mmol/L) during the prolonged exercise

SECONDARY OUTCOMES:
Recovery Interstitial Glucose | 24 hours
  Using CGM to measure recovery glucose levels post-exercise to analyze time in target range, time in hypoglycemia (< 4.0 mmol/L) and time in hyperglycemia (> 10.0 mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Riddell, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No